CLINICAL TRIAL: NCT00187122
Title: Treatment for Newly Diagnosed Patients With Stage III/IV Non-Hodgkin Lymphoma-Study XIII (A Therapeutic Pilot Study)
Brief Title: Treatment for Patients With Stage III or IV Non-Hodgkin Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Raul C. Ribeiro, M.D./Principal Investigator, St.Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHL13
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Lymphoblastic Lymphoma
Keywords: Non-Hodgkin; Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma | interventions — Vincristine; Radiotherapy; Daunorubicin; Asparaginase; Cytarabine; Methotrexate; Mercaptopurine; Etoposide; etoposide phosphate; Cyclophosphamide; Prednisone; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): See Detailed Description section for description of treatment plan.
  Interventions: Drug: Vincristine; Procedure: Radiation Therapy; Drug: Daunomycin; Drug: L-Asparaginase; Drug: Cytarabine; Drug: Methotrexate; Drug: Mercaptopurine; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Prednisone; Drug: Dexamethasone

INTERVENTIONS:
Drug: Vincristine — See Detailed Description section for description of treatment plan.
  Other Names: Oncovin®, Vincasar Pfs®
Procedure: Radiation Therapy — See Detailed Description section for description of treatment plan.
Drug: Daunomycin — See Detailed Description section for description of treatment plan.
  Other Names: Cerubidine®
Drug: L-Asparaginase — See Detailed Description section for description of treatment plan.
  Other Names: Elspar®, Kidrolase®
Drug: Cytarabine — See Detailed Description section for description of treatment plan.
  Other Names: Cytosar-U®
Drug: Methotrexate — See Detailed Description section for description of treatment plan.
  Other Names: Rheumatrex®, TrexallTM
Drug: Mercaptopurine — See Detailed Description section for description of treatment plan.
  Other Names: Purinethol ®
Drug: Etoposide — See Detailed Description section for description of treatment plan.
  Other Names: Toposar®, VePesid®, Etopophos®
Drug: Cyclophosphamide — See Detailed Description section for description of treatment plan.
  Other Names: Cytoxan®, Neosar®
Drug: Prednisone — See Detailed Description section for description of treatment plan.
  Other Names: Deltasone®, Liquid Pred®, Meticorten®, Orasone®
Drug: Dexamethasone — See Detailed Description section for description of treatment plan.
  Other Names: Decadron, Diodex, Hexadrol, Maxidex

SUMMARY:
The main purpose of this study is to determine if it is feasible to administer an intensified, multi-agent chemotherapy regimen for children with stage III and IV non-Hodgkin lymphoma and to find out what the toxicities are.

DETAILED DESCRIPTION:
The overall objective of this research study is to determine the toxicity and feasibility of administration of an intensified, multi-agent chemotherapy regimen for children with stages III and IV non-Hodgkin lymphoma (NHL), lymphoblastic histiotype. The planned pilot therapy includes major modifications of our best previous treatments for patients with T-cell acute lymphoblastic leukemia (ALL) that may improve the disease-free survival of these children and adolescents. Ultimately, it is intended to propose this therapy for further evaluation in the setting of a patient population large enough to evaluate its efficacy.

Secondary objectives are:

* To determine the toxicity of high-dose methotrexate (HDMTX) given prior to the induction/consolidation phase of therapy and of repeated induction treatment (weeks 16-21) in patients with advanced stage NHL, lymphoblastic histiotype.
* To determine the toxicity and feasibility of administration of continuation therapy which include additional drug pairs not used in the St. Jude Total XI-ALL study.
* To estimate the complete response (CR) rate and event-free survival (EFS) in children with stage III/IV lymphoblastic NHL after treatment with this intensified multiagent chemotherapy. Pooling of data from this study with that gained from treatment of patients with T-ALL on the Total XIII and XIII B studies, with appropriate stratification, will facilitate this aim.
* To compare plasma and cerebrospinal fluid concentrations of VP-16 after 1 hour of administration. The data obtained here will be pooled for analysis with that from Total XIII and Total XIII B studies
* To assess serially whether the frequency of specific HPRT mutations in are related to cumulative dose of etoposide, or plasma AUC of etoposide, etoposide catechol, or both
* To assess the degree of bone marrow infiltration at the time of diagnosis and serially during remission using and comparing morphologic, immunologic and molecular methods. In the absence of morphologically detected tumor cells, we will estimate the frequency of minimal residual disease (MRD) during remission using immunologic and molecular methods. The data obtained here will be pooled for analysis with that obtained from T-cell ALL cases treated on Total XIII and Total XIII B ALL studies.
* Because similar studies are being conducted for patients with T-ALL on the Total XIII and Total XIII B ALL studies, we will pool data from the present study with that from T-cell ALL cases treated on Total XIII and Total XIII B ALL studies and correlate detection of lymphoblasts in bone marrow or cerebrospinal fluid (CSF) with subsequent clinical course (complete remission duration).
* To evaluate the sensitivity of neoplastic cells at diagnosis to anticancer drugs. This evaluation will be limited to patients with bone marrow involvement or viable tumor samples at diagnosis. Information obtained from this aim will complement that obtained from patients with T-ALL in the Total XIII and Total XIII B ALL studies.

Details of Treatment Plan:

Pre-Induction Chemotherapy

Methotrexate 200 mg/m2/hr IV push, then 800 mg/m2 IV over 24 hours

Induction

Induction Chemotherapy uses several chemotherapy drugs to kill cancer cells in the body and lasts 6 to 8 weeks.

Prednisone 40 mg/m2/day PO, days 1-29, Vincristine 1.5 mg/m2/week IV, days 1, 8, 15, 22, Daunomycin 25 mg/m2/week IV, days 1, 8, L-asparaginase 10,000 Units/m2 IM days 2, 4, 6, and 8 Etoposide 300 mg/m2 IV Days 22, 25, 29, Cytarabine 300 mg/m2 IV Days 22, 25, 29 For infants less than 12 months of age, Vincristine dosage is 0.05 mg/kg/dose. CNS Therapy

All patients will receive triple IT therapy on days 1, 22, and 43. Patients with known CNS disease will receive additional IT treatments until 2 consecutive CSF studies are normal. Children with cranial nerve palsies will receive local irradiation to the base of the skull.

Consolidation:

HDMTX 2 g/m2 days 44 and 51. Mercaptopurine 75 mg/m2 PO daily, for 14 days. ITMHA will be given into spinal fluid (IT) the day before first HDMTX dose.

Continuation

Continuation: Continuation therapy lasts 120 weeks. The following drugs will be given in different two-drug combinations during this treatment:

Weeks:

1 VP-16 + Cyclo, 2* 6-MP + MTX, 3 MTX + Ara-C, 4 Dex + VCR, 5 VP-16 + Cyclo, 6 6-MP + HDMTX, 7 VP-16 + Ara-C, 8 Dex + VCR 9 VP-16 + Cyclo, 10 6-MP + MTX, 11 MTX + Ara-C, 12 Dex + VCR, 13 VP-16 + Cyclo, 14* 6-MP + HDMTX, 15 VP-16 + Ara-C

IT MHA (MTX, hydrocortisone, Ara-C, dose age dependent, given one day before HDMTX. IT MHA (every 4 weeks) for patients with CNS 2 or 3 status. Reinduction therapy (same as initial induction treatment, except that only one dose of VP-16/ara-C will be given on day 22) will be given from weeks 16 to 21.

Dosages, Schedules and Routes VP-16: 300 mg/m2 IV over 1 hour; once a week, Cyclophosphamide: 300 mg/m2 IV push; once a week, Mercaptopurine (6-MP): 75 mg/m2 PO; daily x 7, Methotrexate (MTX): 40 mg/m2 IM or IV once a week; only IM after CNS radiation, Cytarabine (Ara-C) 300 mg/M2 IV push; once a week, Dexamethasone (Dex): 8 mg/m2 PO; in 3 divided doses daily x 7, Vincristine (VCR) 1.5 mg/m2 IV; once a week (max 2 mg) L-Asparaginase, (L-ASP): 10,000 U/m2 IM; every 4 weeks x 9, HDMTX: 2 g/m2 IV over 2 hours; every 8 weeks x 7 (same leucovorin rescue as used in consolidation phase)

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV Lymphoblastic Lymphoma
* One week or less of prior therapy, only to include steroids, vinca alkaloids, and emergency radiation therapy to the mediastinum in those with severe respiratory.

Exclusion criteria:

* Patients with superior vena cava syndrome, significant compression of the trachea requiring more than 40% oxygen or having significant dyspnea at normal activity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 1993-03; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
To determine toxicity and feasibility of intensified multiagent chemotherapy and high dose methotrexate. | Within first 30 days following pre-induction chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Raul C. Ribeiro, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org